CLINICAL TRIAL: NCT03052218
Title: Evaluation of Pupillometry for CYP2D6 Phenotyping in Children Treated With Tramadol
Acronym: PUPICYP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in recruitment
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Frédérique Rodieux, Dr. Med, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-01936
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Drug Intolerance; Cytochrome P450 CYP2D6 Enzyme Deficiency; Drug Effect
Keywords: children; pain; Cytochrome P450 CYP2D6 genotype; Cytochrome P450 CYP2D6 phenotype; Pupillometry
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm study (Experimental): pupillometry, CYP2D6 genotyping and phenotyping
  Interventions: Device: Pupillometry

INTERVENTIONS:
Device: Pupillometry — Pupillometry performed before administration of tramadol, at T0 and then 1 to twice per hour, during the stay of the patient in the emergency department

SUMMARY:
Pupillometry will be performed before administration of tramadol, at T0 and then 1 to twice per hour in children having received tramadol as a pain killer as part of his/her routine care.

Pupillometry measurement will be correlate to CYP2D6 phenotype and CYP2D6 genetic score

DETAILED DESCRIPTION:
The proposed study is a single-center, observational and prospective study which will be conducted at the Pediatric Emergency Department, Geneva Children's Hospital.

This study will begin in January 2016 and will last one year. 53 patients are planned to be enrolled.

Children receiving oral tramadol as a pain killer at the emergency department, as part of their routine care, will be informed of the current study. Patients willing to participate will be included in the study after signing the inform consent (or respectively his/her parents or legal guardians). A unique oral dose of dextromethorphan (0.15 mg/kg) will be given to the participant for CYP2D6 phenotyping (T0).

Two hours later, capillary whole blood will be sampled to 1) measure the metabolic ratio dextrorphan/dextromethorphan (MRDOR/DEM) in order to determine CYP2D6 phenotype (validated metrics for CYP2D6 phenotyping), 2) measure tramadol and its active metabolite O-desmethyltramadol (M1), and 3) to genotype for CYP2D6. Saliva sample will also be performed to genotype for CYP2D6. Pupillometry will be performed before administration of tramadol, at T0 and then 1 to twice per hour, throughout the patient's stay at the emergency department.

ELIGIBILITY:
Inclusion criteria

* Age 1-15 year at time of inclusion
* Weight ≥ 10 kg
* Treatment with tramadol as a pain killer administrated as part of their routine care
* Parent/Legal guardian has been informed about the study and has signed Informed Consent Form

Exclusion criteria

* Known kidney or liver disease
* Concomitant treatment with inhibitors/inducers of CYP2D6 and CYP3A
* Documented previous adverse reaction to tramadol or dextromethorphan
* Concomitant treatment with any opiate drug and/or any drug with a known impact on pupil size
* Any concomitant condition, which in the opinion of the investigator would preclude a subject's participation in the study

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
pupillometry parameters and CYP2D6 phenotype | 0-6hours after tramadol administration
  Correlation between pupillometry parameters and CYP2D6 phenotype

SECONDARY OUTCOMES:
pupillometry parameters and CYP2D6 genotype | 0-6hours after tramadol administration
  Correlation between pupillometry parameters and CYP2D6 genotype
pupillometry parameters and tramadol concentration | 0-6hours after tramadol administration
  Correlation between pupillometry parameters and blood levels of tramadol and its active metabolite M1

CONTACTS AND LOCATIONS:
Overall Officials: Frederique j Rodieux, MD, Principal Investigator — Division of Clinical Pharmacology and Toxicology Geneva University Hospitals, Geneva, Switzerland
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No